CLINICAL TRIAL: NCT06557863
Title: Reducing Burden in Care Partners of Community-Dwelling Persons With Dementia and Oropharyngeal Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Liron Sinvani, Associate Professor, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24-0196; R61AG079930 (NIH)
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Caregiver Burden; Alzheimer Disease; Dementia; Oropharyngeal Dysphagia
MeSH Terms: conditions — Caregiver Burden; Alzheimer Disease; Dementia; Deglutition Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Control + WeCareToFeedDysphagia (Experimental): Participants receive usual care from their medical team and receive contact information for speech-language pathology follow-up care. Participants will also receive access to the WeCareToFeedDysphagia web tool and receive text message reminders to use the tool.
  Interventions: Behavioral: WeCareToFeedDysphagia web tool
- Enhanced Control (No Intervention): Participants receive usual care from their medical team and receive contact information for speech-language pathology follow-up care.

INTERVENTIONS:
Behavioral: WeCareToFeedDysphagia web tool — The web tool uses written and video content, care-partner testimonials, frequently asked questions, and resource links to provide accurate information (e.g., dysphagia diets), set realistic expectations, identify/support feeding goals (quality of life considerations), acknowledge/support care-partner feelings, and provide competencies/skills for oropharyngeal dysphagia (OD) management.
  Arms: Enhanced Control + WeCareToFeedDysphagia

SUMMARY:
The goal of this clinical trial is to learn if a newly-created website tool, called WeCareToFeedDysphagia, helps to reduce feelings of burden in care partners of patients with Alzheimer's disease and related dementias (AD/ADRD) who were diagnosed with trouble swallowing (oropharyngeal dysphagia). The main questions this first test (pilot) study aims to answer are:

* With the data this pilot study will collect, how do we best measure how strong a relationship is between care partners who use WeCareToFeedDysphagia and reduced feelings of burden (effect size estimates)?
* Is it possible (feasible) to successfully repeat this study in a larger clinical trial with more research participants?

Researchers will compare a group of care partners who have access to the WeCareToFeedDysphagia tool (intervention) to a group of care partners who do not have access to the tool. Both groups will receive contact information for help from a speech language pathologist expert (enhanced usual care).

Participants will:

* be given access to the web tool and receive 3 text message reminders over 3 weeks to use the tool (intervention group only).
* be asked to complete a remote, web-based survey three times: when enrolled in the study, at 1 month following patient leaving the hospital, and at 3 months following patient leaving the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Self identifies as the primary care partner of an older adult patient (patient aged 65 years or older) with Alzheimer's disease and related dementias (AD/ADRD) and oropharyngeal dysphagia (OD) admitted to the Northwell Health medicine service
* Care partner age 18 years or older
* Designated as the legally authorized representative (LAR) or health care proxy (HCP), or designated by the LAR or HCP to participate
* Proficient in English
* Has access to a device (e.g. smartphone, iPad, computer) capable of accessing a web browser

Exclusion Criteria:

* Care partner of patient with a percutaneous feeding tube [i.e. percutaneous endoscopic gastrostomy (PEG) tube, percutaneous endoscopic jejunostomy (PEJ) used exclusively]
* Care partner of patient who will not be discharged to the home or community setting (e.g., home, assisted living, independent living)
* Care partner will not be involved with OD management (e.g. buying or making food, feeding, supervising) after hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Mean Care Partner Burden at 3 Months Post Hospital Discharge | Baseline and 3 months
  Burden will be measured using the Zarit Burden Scale (ZBI-22), a validated measure that assesses 22 statements related to personal strain accompanying caring for another person, which is rated with 5 frequency-related response categories, scored 0 (never) to 4 (nearly always). The total score ranges between 0 and 88 (higher scores indicating higher burden). A score less than 21 has been suggested to indicate care-partner burden. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message. Change will be calculated as the mean value at 3 months minus the mean value at baseline.

SECONDARY OUTCOMES:
Change from Baseline in Mean Care Partner Burden at 1 Month Post Hospital Discharge | Baseline and 1 Month Post Hospital Discharge
  Burden will be measured using the Zarit Burden Scale (ZBI-22), a validated measure that assesses 22 statements related to personal strain accompanying caring for another person, which is rated with 5 frequency-related response categories, scored 0 (never) to 4 (nearly always). The total score ranges between 0 and 88 (higher scores indicating higher burden). A score less than 21 has been suggested to indicate care-partner burden. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message. Change will be calculated as the mean value at 1 month minus the mean value at baseline.
Change from Baseline in Care Partner Quality of Life at 1 Month Post Hospital Discharge | Baseline and 1 Month Post Hospital Discharge
  Care Partner Quality of Life (CarerQol) will be measured using the validated Care-Related Qol-7D. The Care-Related Qol-7D measures well-being (CarerQol-VAS or visual analog scale) and subjective burden. The CarerQol-VAS measures happiness, using endpoints between 'completely unhappy' (0) and 'completely happy' (10). Subjective burden is measured on 7 dimensions (fulfillment, relational problems, mental health, daily activities problems, physical health, and support), and rated as (i) no, (ii) some, and (iii) a lot. The weighted score ranges from 0-100 (worst to best caregiving situation). Higher scores indicate higher quality of life. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message. Change will be calculated as the mean value at 1 month minus the mean value at baseline.
Change from Baseline in Care Partner Quality of Life at 3 Months Post Hospital Discharge | Baseline and 3 Months Post Hospital Discharge
  Care Partner Quality of Life (CarerQol) will be measured using the validated Care-Related Qol-7D. The Care-Related Qol-7D measures well-being (CarerQol-VAS or visual analog scale) and subjective burden. The CarerQol-VAS measures happiness, using endpoints between 'completely unhappy' (0) and 'completely happy' (10). Subjective burden is measured on 7 dimensions (fulfillment, relational problems, mental health, daily activities problems, physical health, and support), and rated as (i) no, (ii) some, and (iii) a lot. The weighted score ranges from 0-100 (worst to best caregiving situation). Higher scores indicate higher quality of life. Outcome measures will be captured through a link to an online questionnaire which will be sent to the care partner's smart phone/device via text message. Change will be calculated as the mean value at 3 months minus the mean value at baseline.
Percent Engagement with the WeCareToFeedDysphagia Tool | 3 Months Post Hospital Discharge
  Engagement with WeCareToFeedDysphagia will be defined as percent of care partners viewing 2 or more pages within the tool. Success will be defined as greater than or equal to 45% of care partners engaging with the tool. Data will be captured via Google Analytics data to assess program usage in the domains of time/date of login, duration of page views, and document downloaded Engagement with the tool will be reported for the intervention arm only.
Percent Consented in Pilot Study | Study completion, up to 1 year
  Percent consented will be calculated as care partners consented over eligible and approached. Success will be defined as greater than or equal to 40% of care partners approached will volunteer to enroll in the study.
Percent Care Partner Attrition at 1 Month Post Hospital Discharge | 1 Month Post Hospital Discharge.
  Percent attrition will be calculated as the total number of consented participants who did not complete the 1 month assessment over the total number of consented participants. Success will be defined as less than or equal to 30% attrition at 1 month post hospital discharge.
Percent Care Partner Attrition at 3 Months Post Hospital Discharge | 3 Months Post Hospital Discharge.
  Percent attrition will be calculated as the total number of consented participants who did not complete the 3 month assessment over the total number of consented participants. Success will be defined as less than or equal to 30% attrition at 3 months post hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Liron Sinvani, MD, Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institutes for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All data which can be sufficiently deidentified to preserve participant confidentiality will be made available via the Open Science Framework (OSF) repository. The goal of all shared data will be to facilitate replication of all primary and secondary, and exploratory study analyses as well as to allow for additional analyses with available data. Data will be redacted according to the safe-harbor method, and effective strategies will be adopted to minimize risk of disclosing a participant's identity. Data will be shared along with documentation of how variables were cleaned, coded, or summarized. In cases where participant-level data could be used to identify individuals, summary data will be presented (e.g. presenting an age category ">85 years old" rather than individual participant age). Information about how summary data was generated will be provided in the data dictionary.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study data and metadata will be available in advance of the first online publication of the primary study outcomes. De-identified data will be stored on OSF indefinitely to allow for continued access.
Access Criteria: Data will be made publicly available
URL: https://osf.io/7t2vy/